CLINICAL TRIAL: NCT01469052
Title: Phase I, Open-Label, Multicenter, Dose-Escalation Study Of The Tyrosine Kinase Inhibitor Of VEGFR-2, AG013736, In Patients With Advanced Solid Tumors
Brief Title: First In Human, Phase 1 Study of AG013736 In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG013736-001; A4060010
Record Dates: First submitted 2011-11-02; First posted 2011-11-10 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental)
  Interventions: Drug: AG-013736
- Cohort 2 (Experimental)
  Interventions: Drug: AG-013736
- Cohort 3 (Experimental)
  Interventions: Drug: AG-013736
- Cohort 4 (Experimental)
  Interventions: Drug: AG-013736
- Cohort 5 (Experimental)
  Interventions: Drug: AG-013736
- Cohort 6 (Experimental)
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — Axitinib continuous oral dosing (10 mg once a day, 10 mg twice a day, 20 mg twice a day or 30 mg twice day) in the fed state
  Arms: Cohort 1
Drug: AG-013736 — Axitinib continuous oral dosing (20 mg twice a day) in the fed state
  Arms: Cohort 2
Drug: AG-013736 — Axitinib continuous oral dosing (5 mg twice a day) in the fed state
  Arms: Cohort 3
Drug: AG-013736 — Axitinib continuous oral dosing (15 mg once a day) in the fed state
  Arms: Cohort 4
Drug: AG-013736 — Axitinib continuous oral dosing (5 mg twice a day) in the fasted state
  Arms: Cohort 5
Drug: AG-013736 — Axitinib continuous oral dosing (2 mg twice a day on the first day of dosing, followed by 5 mg twice a day) in the fasted state
  Arms: Cohort 6

SUMMARY:
The purpose of the study was to characterize the safety of investigational agent AG-013736, in patients with solid tumors in this First In Human trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically or histologically confirmed solid tumor(s) and with at least one measurable disease site
* Patients with adequate bone marrow, liver and kidney function
* Patients with life expectancy of at least 12 weeks

Exclusion Criteria:

* Patients who have received chemotherapy, immunotherapy, radiotherapy or any investigational agent within 4 weeks of study entry
* Patients with have had a major surgical procedure within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-11; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AG013736-001&StudyName=First%20In%20Human%2C%20Phase%201%20Study%20of%20AG013736%20In%20Patients%20With%20Solid%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed: Single dose of axitinib (AG-013736) 10 milligram (mg) tablet orally once daily (QD) followed by 30 mg single dose after 48 hours. Axitinib (AG-013736) 10 mg/ 20 mg/ 30 mg tablet orally twice daily (BID) in fed state continuously in cycles of 4 weeks, up to 8 cycles.
- Cohort 2: Axitinib 20 mg BID, Fed: Axitinib (AG-013736) 20 mg tablet orally BID in fed state continuously in cycles of 4 weeks, up to 8 cycles.
- Cohort 3: Axitinib 5 mg BID, Fed: Axitinib (AG-013736) 5 mg tablet orally BID in fed state continuously in cycles of 4 weeks, up to 8 cycles.
- Cohort 4: Axitinib 15 mg QD, Fed: Axitinib (AG-013736) 15 mg tablet orally QD in fed state continuously in cycles of 4 weeks, up to 8 cycles.
- Cohort 5: Axitinib 5 mg BID, Fasted: Axitinib (AG-013736) 5 mg tablet orally BID in fasted state continuously in cycles of 4 weeks, up to 8 cycles.
- Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted: Axitinib (AG-013736) 2 mg tablet orally BID on the first day of dosing followed by 5 mg BID in fasted state continuously in cycles of 4 weeks, up to 8 cycles.
Period: Overall Study
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Started | 6 | 4 | 6 | 6 | 8 | 6
Completed | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 6 | 4 | 6 | 5 | 8 | 6
Not completed — Adverse Event | 2 | 3 | 0 | 2 | 0 | 1
Not completed — Progressive disease | 3 | 0 | 5 | 3 | 7 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Moved to rollover protocol | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed: Single dose of axitinib (AG-013736) 10 mg tablet orally QD followed by 30 mg single dose after 48 hours. Axitinib (AG-013736) 10 mg/ 20 mg/ 30 mg tablet orally BID in fed state continuously in cycles of 4 weeks, up to 8 cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted | Total
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6 | 36
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.83 (8.75) | 58.50 (4.80) | 55.00 (7.27) | 56.00 (9.44) | 54.88 (7.95) | 64.17 (10.01) | 56.86 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 2 | 5 | 3 | 20
  Male | 2 | 0 | 4 | 4 | 3 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the dose level at which "no more than 1 of 6 participants experience dose-limiting toxicity (DLT) following de-escalation from the maximum administered dose (MAD)." DLT includes grade (Gr) 2 or greater gastrointestinal toxicities, Gr 3 anemia, nonhematological toxicities (excluding nausea, vomiting, and diarrhea) or Gr 4 neutropenia, thrombocytopenia and inability to resume axitinib (AG-013736) dosing within 14 days of stopping due to treatment related toxicity.
Time Frame: Baseline up to Day 28
Population: Analysis population included all enrolled participants who received at least one dose of the study drug.
Measure: Number; unit: mg BID
Groups:
- All Treated Participants: All participants of Cohorts 1 to 6 received oral doses of axitinib (AG-013736) (10 mg and 15 mg, QD; 2 mg, 5 mg, 10 mg, 20 mg and 30 mg, BID) tablet in fed or fasted state in cycles of 4 weeks, up to 8 cycles.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 36
mg BID | 5

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hours (hrs) post-dose on Day (D) 1 and 15 of Cycle (C) 1 and Day 29 (Day 1 of Cycle 2); pre-dose on Day 43 (Day 15 of Cycle 2) and Day 57 (Day 1 of Cycle 3)
Population: Analysis population included all enrolled participants who received at least one dose of the study drug.'n' signifies those participants evaluated for this measure at specific time point for each cohort respectively.
Measure: Geometric Mean (Standard Deviation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6
Nanogram/milliliter (ng/mL)
  Day 1 (n= 6, 4, 6, 5, 8, 6) | 144.48 (73.90) | 97.81 (89.96) | 20.71 (9.48) | 88.16 (84.93) | 22.21 (34.88) | 19.75 (17.95)
  Day 15 (n= 6, 3, 5, 6, 6, 6) | 130.91 (60.23) | 94.75 (110.81) | 28.68 (8.33) | 67.08 (42.50) | 51.82 (31.21) | 52.24 (53.87)
  Day 29 (n= 4, 3, 5, 5, 7, 6) | 76.25 (67.86) | 69.14 (103.14) | 26.44 (17.28) | 60.11 (103.76) | 43.28 (41.41) | 60.48 (29.10)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 1 and 15 of Cycle 1 and Day 29 (Day 1 of Cycle 2); pre-dose on Day 43 (Day 15 of Cycle 2) and Day 57 (Day 1 of Cycle 3)
Population: Analysis population included all enrolled participants who received at least one dose of the study drug. 'n' signifies those participants evaluated for this measure at specific time point for each cohort respectively.
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6
hr
  Day 1 (n= 6, 4, 6, 5, 8, 6) | 2.00 [1.00 to 4.00] | 4.04 [2.00 to 8.03] | 4.00 [1.00 to 4.08] | 2.05 [1.98 to 4.00] | 1.52 [0.50 to 4.00] | 1.01 [1.00 to 4.00]
  Day 15 (n= 6, 3, 5, 6, 6, 6) | 3.00 [1.00 to 4.00] | 3.95 [2.08 to 4.05] | 2.00 [1.00 to 4.22] | 4.00 [2.00 to 11.83] | 1.01 [0.98 to 2.03] | 1.51 [0.98 to 4.00]
  Day 29 (n= 4, 3, 5, 5, 7, 6) | 3.44 [0.00 to 4.03] | 4.13 [1.00 to 11.98] | 2.00 [1.00 to 4.00] | 3.50 [2.00 to 8.97] | 1.00 [0.50 to 4.02] | 2.01 [0.98 to 4.00]

4. Secondary Outcome: Area Under the Curve From Time Zero to 12 Hours [AUC (0-12)]
Description: AUC (0-12)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-12).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6
ng*hr/mL
  Day 1 (n= 6, 4, 6, 5, 8, 6) | 692.47 [363.89 to 1317.76] | 564.56 [100.47 to 3172.37] | 88.62 [60.05 to 130.80] | 473.26 [162.59 to 1377.58] | 68.73 [29.84 to 158.34] | 61.92 [19.33 to 198.31]
  Day 15 (n= 6, 3, 5, 6, 6, 6) | 793.89 [372.39 to 1692.48] | 485.52 [15.97 to 14760.66] | 130.57 [77.24 to 220.72] | 380.56 [161.49 to 896.80] | 126.25 [50.65 to 314.70] | 218.05 [81.21 to 585.47]
  Day 29 (n= 4, 3, 5, 5, 7, 6) | 456.53 [98.07 to 2125.11] | 441.50 [19.51 to 9989.18] | 144.13 [66.74 to 311.24] | 377.86 [104.98 to 1360.02] | 126.08 [55.72 to 285.29] | 253.45 [127.21 to 504.96]

5. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hr (L/hr)
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6
Liter/hr (L/hr)
  Day 1 (n= 6, 4, 6, 5, 8, 6) | 19.80 [9.14 to 42.87] | 30.82 [5.00 to 189.99] | 53.17 [35.99 to 78.55] | 29.04 [10.34 to 81.59] | 71.82 [31.26 to 165.04] | 30.27 [8.95 to 102.37]
  Day 15 (n= 6, 3, 5, 6, 6, 6) | 18.82 [8.90 to 39.78] | 32.69 [2.80 to 381.94] | 38.29 [22.65 to 64.73] | 30.61 [11.26 to 83.23] | 39.05 [15.38 to 99.13] | 22.93 [8.54 to 61.57]
  Day 29 (n= 4, 2, 5, 5, 7, 6) | 27.32 [8.35 to 89.42] | 18.82 [0.00 to NA] — The upper limit of Confidence interval was not estimable since only 2 participants were evaluable. | 34.69 [16.06 to 74.91] | 31.07 [7.11 to 135.74] | 38.51 [16.66 to 89.02] | 19.73 [9.90 to 39.31]

6. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: Axitinib (10 mg QD + 10 mg/20mg/30mg BID), Fed | Cohort 2: Axitinib 20 mg BID, Fed | Cohort 3: Axitinib 5 mg BID, Fed | Cohort 4: Axitinib 15 mg QD, Fed | Cohort 5: Axitinib 5 mg BID, Fasted | Cohort 6: Axitinib 2 mg + 5 mg BID, Fasted
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 8 | 6
hr
  Day 1 (n= 6, 3, 5, 5, 5, 4) | 3.09 (1.00) | 3.29 (1.86) | 2.31 (0.64) | 3.08 (0.97) | 1.86 (0.44) | 3.77 (1.60)
  Day 15 (n= 5, 3, 5, 4, 5, 6) | 5.20 (3.12) | 3.17 (1.71) | 2.22 (0.34) | 2.48 (0.68) | 2.01 (1.23) | 5.78 (6.33)
  Day 29 (n= 3, 2, 5, 3, 6, 6) | 6.11 (4.23) | 3.94 (2.65) | 2.78 (0.80) | 2.16 (0.79) | 3.03 (0.74) | 3.33 (0.90)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) in Fed State Versus Overnight Fasting
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 29 (Day 1 of Cycle 2) and Day 30 (Day 2 of Cycle 2)
Population: The actual mean values were not reported in the fed and fasted state because the food effect evaluation was conducted across different dose groups and hence it was not appropriate to report overall mean values in different doses as PK parameters change with dose.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Fed State: Axitinib (AG-013736) tablet 5 mg BID, 15 mg QD and 20 mg BID were administered orally in fed state in cycles of 4 weeks, up to 8 cycles.
- Fasted State: Axitinib (AG-013736) tablet 5 mg BID, 15 mg QD and 20 mg BID were administered orally in fasted state in cycles of 4 weeks, up to 8 cycles.
Arm/Group | Fed State | Fasted State
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) in Fed State Versus Overnight Fasting
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 29 (Day 1 of Cycle 2) and Day 30 (Day 2 of Cycle 2)
Population: as for outcome 7
Measure: Mean (90% Confidence Interval); unit: hr
Arm/Group | Fed State | Fasted State
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC (0-24)] in Fed State Versus Overnight Fasting
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 29 (Day 1 of Cycle 2) and Day 30 (Day 2 of Cycle 2)
Population: as for outcome 7
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Arm/Group | Fed State | Fasted State
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Apparent Oral Clearance (CL/F) in Fed State Versus Overnight Fasting
Description: as for outcome 5
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 29 (Day 1 of Cycle 2) and Day 30 (Day 2 of Cycle 2)
Population: as for outcome 7
Measure: Geometric Mean (90% Confidence Interval); unit: L/hr
Arm/Group | Fed State | Fasted State
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Plasma Decay Half-Life (t1/2) in Fed State Versus Overnight Fasting
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, and 12 hrs post-dose on Day 29 (Day 1 of Cycle 2) and Day 30 (Day 2 of Cycle 2)
Population: as for outcome 7
Measure: Geometric Mean (90% Confidence Interval); unit: hr
Arm/Group | Fed State | Fasted State
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | All Treated Participants
Serious Adverse Events (participants affected / at risk) | 12/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (N=36)
Dysphagia (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Eye pain (Eye disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Convulsion (Nervous system disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (N=36)
Anaemia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 3
Retching (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 4
Chest pain (General disorders) | 2
Fatigue (General disorders) | 16
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 3
Thirst (General disorders) | 2
Infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 18
Dysphagia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Oral discomfort (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.